CLINICAL TRIAL: NCT06705894
Title: Risk of Respiratory Complications Following Gastrointestinal Endoscopy Under Monitored Anesthesia Care: A Prospective Cohort Study
Brief Title: Risk of Respiratory Complications Following Gastrointestinal Endoscopy Under Monitored Anesthesia Care
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jixiangyu, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYEC2024-218
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-04

CONDITIONS: Pneumonia, Aspiration
Keywords: Gastrointestinal endoscopy; Respiratory complications; Sedation
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- M group: Gratrointestinal endoscopy is undergone with moderate sedation.
- D/G group: Gratrointestinal endoscopy is undergone without deep sedation/general anesthsia.

SUMMARY:
The purpose of this study is to investigate the incidence of respiratory complications after gastroenteroscopy, and establish a Logistic regression model to analyze the related risk factors of respiratory complications.

DETAILED DESCRIPTION:
Gastrointestinal endoscopy is currently the most widely used and reliable technique for diagnosing digestive tract diseases.With the increasing need for pain relief and the improvement of anesthesiology technology, more and more patients prefer to undergo gastroenteroscopy under sedation or anesthesia.The painless technique of gastroenteroscopy is an anesthetic method , and like other anesthesia techniques, it brings risks as well as comfort.However, current studies mainly focus on respiratory and circulation-related adverse events during the examination , while little attention is paid to delayed respiratory complications after examination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Qualified gastrointestinal tract preparation in strict accordance with the preparation requirements related to gastroenteroscopy;

Exclusion Criteria:

1. Patients with respiratory system symptoms or history before surgery;
2. Patients in need of a tracheal intubation;
3. Refuse follow-up;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population undergoing gastrointestinal endoscopy examination at Qingdao University Affiliated Hospital from December 2024 to February 2025.
Sampling Method: Non-Probability Sample
Enrollment: 10313 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative cough | 24 hours after surgery
  The investigator needs to use NRS scores to evaluate the severity of the cough, if patients develop a new cough after surgery.The score from 0 (no) to 10 (extremely serious).Duration and treatment are also required to be recorded.
Postoperative fever | 24 hours after surgery
  The investigator needs to record the patient's maximum body temperature. Duration and treatment are also required to be recorded.
Short of breath | 24 hours after surgery
  The investigator needs to use mMRC questionnaire to evaluate the severity of SOB.Duration and treatment are also required to be recorded.

SECONDARY OUTCOMES:
Adverse events during surgery | During surgery
  Adverse events such as coughing, reflux aspiration, laryngeal spasm, and hypotension need to be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shangdong, China